CLINICAL TRIAL: NCT00468351
Title: Intravitreal Bevacizumab Versus Intravitreal Triamcinolone Acetonide for Refractory Diabetic Macular Edema
Brief Title: Intravitreal Triamcinolone Acetonide Versus Intravitreal Bevacizumab for Refractory Diabetic Macular Edema (IBEME Study)
Acronym: IBEME
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 154342005
Record Dates: First submitted 2007-05-01; First posted 2007-05-02 (Estimated); Last update posted 2007-05-02 (Estimated); Status verified 2007-04

CONDITIONS: Diabetic Macular Edema
Keywords: bevacizumab; diabetes; intravitreal; macular edema; triamcinolone; VEGF
MeSH Terms: conditions — Diabetes Mellitus; Macular Edema | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Intravitreal Injection of 1,5 mg of bevacizumab
Procedure: Intravitreal injection of 4 mg of Triamcinolone acetonide

SUMMARY:
Intravitreal triamcinolone has been effective for central macular thickness reduction and concomitant visual acuity improvement in patients with diabetic macular edema (DME). VEGF is a very effective inducer of permeability, being 50.000 times more potent than histamine, and may exert its effect on retinal vascular permeability by altering tight-junctions proteins, such as occluding and VE-cadherin. Based on these principles, there is a rationale for anti-VEGF agents treatment of increased retinal capillary permeability conditions, such as diabetic macular edema. Therefore, we conducted a randomized, prospective study to compare the efficacy and safety of intravitreal triamcinolone acetonide and intravitreal bevacizumab injection for refractory diffuse DME.

ELIGIBILITY:
Inclusion Criteria:

* Refractory diffuse DME (defined herein as clinically significant DME [by biomicroscopic evaluation] unresponsive to focal laser photocoagulation [performed at least 3 months before evaluation] and generalized breakdown of the inner blood-retina barrier with diffuse fluorescein leakage involving the foveal center and most of the macular area on fluorescein angiography),
* Snellen logarithm of minimum angle of resolution (LogMAR) BCVA equivalent of 20/40 or worse, and 3) central macular thickness (CMT) greater than 300µm on optical coherence tomography (OCT)

Exclusion Criteria:

* Aphakic or pseudophakic eyes,
* Glycosylated hemoglobin (Hb A1C) rate above 10%,
* History of glaucoma or ocular hypertension,
* Loss of vision as a result of other causes,
* Systemic corticoid therapy,.
* History of thromboembolic event (including myocardial infarction or cerebral vascular accident);
* Major surgery within the prior 6 months or planned within the next 28 days;
* Uncontrolled hypertension (according to guidelines of the seventh report of the joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure [JNC-7]);16
* Known coagulation abnormalities or current use of anticoagulative medication other than aspirin;
* Severe systemic disease; or
* Any condition affecting follow-up or documentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-04; Study Completion 2007-04

PRIMARY OUTCOMES:
Central Macular Thickness, Best Corrected Visual Acuity | six months

SECONDARY OUTCOMES:
Intraocular pressure; lens status | six months

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Jorge, MD, PhD, Study Chair — HCFMRP-USP; Rogério A Costa, MD, PhD, Study Director — Retina Diagnostic and Treatment Division, Hospital de Olhos de Araraquara, Araraquara; Rodrigo Jorge, MD, PhD, Principal Investigator — HCFMRP-USP
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Background] Arevalo JF, Fromow-Guerra J, Quiroz-Mercado H, Sanchez JG, Wu L, Maia M, Berrocal MH, Solis-Vivanco A, Farah ME; Pan-American Collaborative Retina Study Group. Primary intravitreal bevacizumab (Avastin) for diabetic macular edema: results from the Pan-American Collaborative Retina Study Group at 6-month follow-up. Ophthalmology. 2007 Apr;114(4):743-50. doi: 10.1016/j.ophtha.2006.12.028. PMID 17398322
- [Background] Bonini-Filho MA, Jorge R, Barbosa JC, Calucci D, Cardillo JA, Costa RA. Intravitreal injection versus sub-Tenon's infusion of triamcinolone acetonide for refractory diabetic macular edema: a randomized clinical trial. Invest Ophthalmol Vis Sci. 2005 Oct;46(10):3845-9. doi: 10.1167/iovs.05-0297. PMID 16186372
- [Background] Costa RA, Jorge R, Calucci D, Melo LA Jr, Cardillo JA, Scott IU. Intravitreal bevacizumab (avastin) for central and hemicentral retinal vein occlusions: IBeVO study. Retina. 2007 Feb;27(2):141-9. doi: 10.1097/IAE.0b013e31802eff83. PMID 17290194
- [Background] Jorge R, Costa RA, Calucci D, Cintra LP, Scott IU. Intravitreal bevacizumab (Avastin) for persistent new vessels in diabetic retinopathy (IBEPE study). Retina. 2006 Nov-Dec;26(9):1006-13. doi: 10.1097/01.iae.0000246884.76018.63. PMID 17151487
- [Background] Costa RA, Jorge R, Calucci D, Cardillo JA, Melo LA Jr, Scott IU. Intravitreal bevacizumab for choroidal neovascularization caused by AMD (IBeNA Study): results of a phase 1 dose-escalation study. Invest Ophthalmol Vis Sci. 2006 Oct;47(10):4569-78. doi: 10.1167/iovs.06-0433. PMID 17003454
- [Background] Audren F, Lecleire-Collet A, Erginay A, Haouchine B, Benosman R, Bergmann JF, Gaudric A, Massin P. Intravitreal triamcinolone acetonide for diffuse diabetic macular edema: phase 2 trial comparing 4 mg vs 2 mg. Am J Ophthalmol. 2006 Nov;142(5):794-99. doi: 10.1016/j.ajo.2006.06.011. Epub 2006 Sep 15. PMID 16978576
- [Background] Chun DW, Heier JS, Topping TM, Duker JS, Bankert JM. A pilot study of multiple intravitreal injections of ranibizumab in patients with center-involving clinically significant diabetic macular edema. Ophthalmology. 2006 Oct;113(10):1706-12. doi: 10.1016/j.ophtha.2006.04.033. PMID 17011952
- [Background] Cunningham ET Jr, Adamis AP, Altaweel M, Aiello LP, Bressler NM, D'Amico DJ, Goldbaum M, Guyer DR, Katz B, Patel M, Schwartz SD; Macugen Diabetic Retinopathy Study Group. A phase II randomized double-masked trial of pegaptanib, an anti-vascular endothelial growth factor aptamer, for diabetic macular edema. Ophthalmology. 2005 Oct;112(10):1747-57. doi: 10.1016/j.ophtha.2005.06.007. PMID 16154196
- [Background] Haritoglou C, Kook D, Neubauer A, Wolf A, Priglinger S, Strauss R, Gandorfer A, Ulbig M, Kampik A. Intravitreal bevacizumab (Avastin) therapy for persistent diffuse diabetic macular edema. Retina. 2006 Nov-Dec;26(9):999-1005. doi: 10.1097/01.iae.0000247165.38655.bf. PMID 17151486
- [Derived] Folgosa MS, Messias A, Takata C, Costa RA, Scott IU, Jorge R. Single intravitreal injection of triamcinolone combined with bevacizumab for the treatment of diffuse diabetic macular oedema refractory to grid photocoagulation. Acta Ophthalmol. 2010 Nov;88(7):e297-8. doi: 10.1111/j.1755-3768.2009.01721.x. No abstract available. PMID 19906082